CLINICAL TRIAL: NCT02848690
Title: The Effectiveness of an Educational Intervention for Sodium Restriction in Patients With Hypertension: Study Protocol for a Randomized Controlled Trial
Brief Title: Educational Intervention for Sodium Restriction in Patients With Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150496
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension,
Keywords: Sodium restriction; Dietary sodium restriction questionnaire (DSRQ); Low-sodium diet; Adherence; Educational intervention
MeSH Terms: conditions — Hypertension | interventions — Early Intervention, Educational; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention Group (Experimental): Participants assigned to the educational intervention group will have dietitian consultation to receive a dietary planning based on diet rich of fruits, vegetables, low fat, low processed foods and high nonfat dairy. During six months they will have monthly dietitian appointments including educational sessions to stimulate sodium restriction and enhance to follow the dietary planning. Each 15 days they will be contacted by phone to reinforce adherence to sodium restriction diet.
  Interventions: Behavioral: Educational Intervention
- Usual Care Intervention Group (Sham Comparator): Participants assigned to the control group will have a dietitian consultation receiving general recommendations for hypertension, such as increasing the consumption of fruits and vegetables, reducing salt intake, avoiding processed and high-sodium foods, reducing body weight if BMI> 25Kg/m2 and limiting consumption of alcoholic beverages. They will be provided with an explanatory folder about hypertension. During six months, participants assigned to the control group will be monitored in monthly visits to the dietitian without modifying their usual care
  Interventions: Other: Usual Care Intervention Group

INTERVENTIONS:
Behavioral: Educational Intervention — The educational intervention sessions will be conducted face-to-face, one hour-long and with the aim to encourage and motivate the low-sodium diet adherence. The dietitian's approaches will provide individual skills to achieve the goals (sodium restriction), developing changes in behavior and monitoring the progress towards the skills needed to reduce patient's barriers and difficulties for sodium restricted diet adherence.
  Other Names: Intervention Group
  Arms: Educational Intervention Group
Other: Usual Care Intervention Group — Participants assigned to the control group will have a dietitian consultation receiving general recommendations for hypertension, such as increasing the consumption of fruits and vegetables, reducing salt intake, avoiding processed and high-sodium foods, reducing body weight if BMI> 25Kg/m2 and limiting consumption of alcoholic beverages. They will be provided with an explanatory folder about hypertension. During six months, participants assigned to the control group will be monitored in monthly visits to the dietitian without modifying their usual care
  Other Names: Control Group
  Arms: Usual Care Intervention Group

SUMMARY:
This parallel, randomized clinical trial will include 120 participants. They will be allocated to a sodium restriction educational intervention or usual care groups. The educational intervention will be planned based on the DSRQ application and sessions will be conducted once a month for the period of six months. Both spot urine collection to estimate sodium intake and the DSRQ will be applied at the baseline, in the eighth week and at the end of the follow-up. Blood sample and 24-hour ambulatory blood pressure monitoring (ABPM) will be conducted at the beginning and at the end of the follow-up. Anthropometric measurements, blood pressure measurement and 24-hour food recall will be collected during follow-up.

DETAILED DESCRIPTION:
This parallel, randomized clinical trial will include 120 participants. They will be allocated to a sodium restriction educational intervention or usual care groups. The educational intervention will be planned based on the DSRQ application and sessions will be conducted once a month for the period of six months. Both spot urine collection to estimate sodium intake and the DSRQ will be applied at the baseline, in the eighth week and at the end of the follow-up. Blood sample and 24-hour ambulatory blood pressure monitoring (ABPM) will be conducted at the beginning and at the end of the follow-up. Anthropometric measurements, blood pressure measurement and 24-hour food recall will be collected during follow-up. The study 'The effectiveness of an educational intervention to sodium restriction in patients with hypertension' is based on the results of the DSRQ application, whose objective is to evaluate aspects related to non-adherence to the recommendation of a low-sodium diet, identifying adherence barriers and facilitators, contributing to the planning of interventions for improving the adoption of a low-sodium diet and, consequently, better hypertension control.

ELIGIBILITY:
Inclusion Criteria:

* female and male individuals, ageing from 40 to 80 years old, in treatment and monitored at the hypertensive outpatient department of HCPA. Participants must not have been monitored by a nutritionist or followed a nutritional orientation for over than six months

Exclusion Criteria:

* pregnancy or lactating; gastrointestinal tract disease; inflammatory disease; chemotherapy treatment; diabetes diagnosis; incapacity to follow an interview and/or to participate in the intervention program without the need of a third party involvement

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline, after 8 weeks and 6 months in Dietary Sodium Restriction Questionnaire (DSRQ) score | 6 months

SECONDARY OUTCOMES:
Questionnaire sensitivity and specificity by the comparison of Dietary Sodium Restriction Questionnaire (DSRQ) scores to urinary sodium values | 6 months
Changes from baseline, after 8 weeks and 6 months in urinary sodium values | 6 months
Changes from baseline, after 8 weeks and 6 months in blood pressure mean assessed by ABPM | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leila Moreira, MD PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Leila Beltrami Moreira, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Result] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Result] Appel LJ, Champagne CM, Harsha DW, Cooper LS, Obarzanek E, Elmer PJ, Stevens VJ, Vollmer WM, Lin PH, Svetkey LP, Stedman SW, Young DR; Writing Group of the PREMIER Collaborative Research Group. Effects of comprehensive lifestyle modification on blood pressure control: main results of the PREMIER clinical trial. JAMA. 2003 Apr 23-30;289(16):2083-93. doi: 10.1001/jama.289.16.2083. PMID 12709466
- [Result] He FJ, MacGregor GA. Effect of longer-term modest salt reduction on blood pressure. Cochrane Database Syst Rev. 2004;(3):CD004937. doi: 10.1002/14651858.CD004937. PMID 15266549
- [Result] Aucott L, Rothnie H, McIntyre L, Thapa M, Waweru C, Gray D. Long-term weight loss from lifestyle intervention benefits blood pressure?: a systematic review. Hypertension. 2009 Oct;54(4):756-62. doi: 10.1161/HYPERTENSIONAHA.109.135178. Epub 2009 Aug 24. PMID 19704106
- [Result] Whelton SP, Chin A, Xin X, He J. Effect of aerobic exercise on blood pressure: a meta-analysis of randomized, controlled trials. Ann Intern Med. 2002 Apr 2;136(7):493-503. doi: 10.7326/0003-4819-136-7-200204020-00006. PMID 11926784
- [Result] Ajani UA, Dunbar SB, Ford ES, Mokdad AH, Mensah GA. Sodium intake among people with normal and high blood pressure. Am J Prev Med. 2005 Dec;29(5 Suppl 1):63-7. doi: 10.1016/j.amepre.2005.07.008. PMID 16389128
- [Result] Reinivuo H, Valsta LM, Laatikainen T, Tuomilehto J, Pietinen P. Sodium in the Finnish diet: II trends in dietary sodium intake and comparison between intake and 24-h excretion of sodium. Eur J Clin Nutr. 2006 Oct;60(10):1160-7. doi: 10.1038/sj.ejcn.1602431. Epub 2006 Apr 26. PMID 16639417
- [Result] Ferreira-Sae MC, Gallani MC, Nadruz W, Rodrigues RC, Franchini KG, Cabral PC, Sales ML. Reliability and validity of a semi-quantitative FFQ for sodium intake in low-income and low-literacy Brazilian hypertensive subjects. Public Health Nutr. 2009 Nov;12(11):2168-73. doi: 10.1017/S1368980009005825. Epub 2009 May 28. PMID 19476677
- [Result] Cornelio ME, Gallani MC, Godin G, Rodrigues RC, Mendes RD, Nadruz Junior W. Development and reliability of an instrument to measure psychosocial determinants of salt consumption among hypertensive patients. Rev Lat Am Enfermagem. 2009 Sep-Oct;17(5):701-7. doi: 10.1590/s0104-11692009000500017. PMID 19967221
- [Result] Polonia J, Martins L. A comprehensive review on salt and health and current experience of worldwide salt reduction programmes. J Hum Hypertens. 2009 Nov;23(11):771-2. doi: 10.1038/jhh.2009.64. Epub 2009 Sep 3. No abstract available. PMID 19727126
- [Result] Appel LJ, Frohlich ED, Hall JE, Pearson TA, Sacco RL, Seals DR, Sacks FM, Smith SC Jr, Vafiadis DK, Van Horn LV. The importance of population-wide sodium reduction as a means to prevent cardiovascular disease and stroke: a call to action from the American Heart Association. Circulation. 2011 Mar 15;123(10):1138-43. doi: 10.1161/CIR.0b013e31820d0793. Epub 2011 Jan 13. No abstract available. PMID 21233236
- [Result] Evers SE, Bass M, Donner A, McWhinney IR. Lack of impact of salt restriction advice on hypertensive patients. Prev Med. 1987 Mar;16(2):213-20. doi: 10.1016/0091-7435(87)90085-5. PMID 3588562
- [Result] Cornelio ME, Gallani MC, Godin G, Rodrigues RC, Nadruz W Jr, Mendez RD. Behavioural determinants of salt consumption among hypertensive individuals. J Hum Nutr Diet. 2012 Aug;25(4):334-44. doi: 10.1111/j.1365-277X.2012.01238.x. Epub 2012 Mar 2. PMID 22380701
- [Result] Adams SO, Maller O, Cardello AV. Consumer acceptance of foods lower in sodium. J Am Diet Assoc. 1995 Apr;95(4):447-53. doi: 10.1016/S0002-8223(95)00120-4. PMID 7699187
- [Result] Mattes RD. The taste for salt in humans. Am J Clin Nutr. 1997 Feb;65(2 Suppl):692S-697S. doi: 10.1093/ajcn/65.2.692S. PMID 9022567
- [Result] Kumanyika SK, Hebert PR, Cutler JA, Lasser VI, Sugars CP, Steffen-Batey L, Brewer AA, Cameron M, Shepek LD, Cook NR, et al. Feasibility and efficacy of sodium reduction in the Trials of Hypertension Prevention, phase I. Trials of Hypertension Prevention Collaborative Research Group. Hypertension. 1993 Oct;22(4):502-12. doi: 10.1161/01.hyp.22.4.502. PMID 8406655
- [Result] Kumanyika SK, Cook NR, Cutler JA, Belden L, Brewer A, Cohen JD, Hebert PR, Lasser VI, Raines J, Raczynski J, Shepek L, Diller L, Whelton PK, Yamamoto M; Trials of Hypertension Prevention Collaborative Research Group. Sodium reduction for hypertension prevention in overweight adults: further results from the Trials of Hypertension Prevention Phase II. J Hum Hypertens. 2005 Jan;19(1):33-45. doi: 10.1038/sj.jhh.1001774. PMID 15372064
- [Result] Welsh D, Lennie TA, Marcinek R, Biddle MJ, Abshire D, Bentley B, Moser DK. Low-sodium diet self-management intervention in heart failure: pilot study results. Eur J Cardiovasc Nurs. 2013 Feb;12(1):87-95. doi: 10.1177/1474515111435604. Epub 2012 Apr 4. PMID 22492785
- [Result] d'Almeida KS, Souza GC, Rabelo ER. Cross-cultural adaptation into Brazilian portuguese of the Dietary Sodium Restriction Questionnaire (DSRQ). Arq Bras Cardiol. 2012 Jan;98(1):70-5. doi: 10.1590/s0066-782x2011005000122. Epub 2011 Dec 15. English, Portuguese, Spanish. PMID 22159403
- [Result] d'Almeida KS, Souza GC, Rabelo-Silva ER. Validity and reliability of the Dietary Sodium Restriction Questionnaire (DSRQ). Nutr Hosp. 2013 Sep-Oct;28(5):1702-9. doi: 10.3305/nh.2013.28.5.6679. PMID 24160236
- [Result] Bentley B, Lennie TA, Biddle M, Chung ML, Moser DK. Demonstration of psychometric soundness of the Dietary Sodium Restriction Questionnaire in patients with heart failure. Heart Lung. 2009 Mar-Apr;38(2):121-8. doi: 10.1016/j.hrtlng.2008.05.006. Epub 2008 Aug 28. PMID 19254630
- [Derived] Rodrigues MP, Dos Santos LKJ, Fuchs FD, Fuchs SC, Moreira LB. The effectiveness of an educational intervention for sodium restriction in patients with hypertension: study protocol for a randomized controlled trial. Trials. 2017 Jul 21;18(1):347. doi: 10.1186/s13063-017-2091-4. PMID 28732546